CLINICAL TRIAL: NCT04256174
Title: A Phase 1, Randomized, Two-Part, Double-Blind, Placebo-Controlled, Dose-Escalation, Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of AK120 in Healthy Subjects and Subjects With Moderate- to- Severe Atopic Dermatitis
Brief Title: A Study of AK120 (IL-4Rα) in Healthy Subjects and Subjects With Moderate- to- Severe Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akesobio Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Akeso (Industry)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: AK120-101
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Part 1:15mg cohort (Experimental): Single dose of 15mg AK120 or placebo is administered subcutaneously to healthy subjects.
  Interventions: Drug: AK120 or placebo- Part 1- Cohort 1
- Part 1: 50mg cohort (Experimental): Single dose of 50mg AK120 or placebo is administered subcutaneously to healthy subjects.
  Interventions: Drug: AK120 or placebo- Part 1- Cohort 2
- Part 1: 150mg cohort (Experimental): Single dose of 150mg AK120 or placebo is administered subcutaneously to healthy subjects.
  Interventions: Drug: AK120 or placebo- Part 1- Cohort 3
- Part 1: 300 mg cohort (Experimental): Single dose of 300mg AK120 or placebo is administered subcutaneously to healthy subjects.
  Interventions: Drug: AK120 or placebo- Part 1- Cohort 4
- Part 1: 600 mg cohort (Experimental): Single dose of 600mg AK120 or placebo is administered subcutaneously to healthy subjects.
  Interventions: Drug: AK120 or placebo- Part 1- Cohort 5
- Part 2: low dose cohort (Experimental): Multiple low doses of AK120 or placebo are administered subcutaneously to subjects with moderate- to- severe atopic dermatitis.
  Interventions: Drug: AK120 or placebo- Part 2- Cohort 1
- Part 2: medium dose cohort (Experimental): Multiple medium doses of AK120 or placebo are administered subcutaneously to subjects with moderate- to- severe atopic dermatitis.
  Interventions: Drug: AK120 or placebo- Part 2- Cohort 2
- Part 2: high dose cohort (Experimental): Multiple high doses of AK120 or placebo are administered subcutaneously to subjects with moderate- to- severe atopic dermatitis.
  Interventions: Drug: AK120 or placebo- Part 2- Cohort 3
- Part 2: Loading dose cohort (Experimental): A loading dose followed by multiple high doses of AK120 or placebo are administered subcutaneously to subjects with moderate- to- severe atopic dermatitis.
  Interventions: Drug: AK120 or placebo- Part 2- Cohort 4

INTERVENTIONS:
Drug: AK120 or placebo- Part 1- Cohort 1 — Single dose of 15mg AK120 or placebo is administered subcutaneously to healthy subjects
  Arms: Part 1:15mg cohort
Drug: AK120 or placebo- Part 1- Cohort 2 — Single dose of 50mg AK120 or placebo is administered subcutaneously to healthy subjects
  Arms: Part 1: 50mg cohort
Drug: AK120 or placebo- Part 1- Cohort 3 — Single dose of 150mg AK120 or placebo is administered subcutaneously to healthy subjects
  Arms: Part 1: 150mg cohort
Drug: AK120 or placebo- Part 1- Cohort 4 — Single dose of 300mg AK120 or placebo is administered subcutaneously to healthy subjects
  Arms: Part 1: 300 mg cohort
Drug: AK120 or placebo- Part 1- Cohort 5 — Single dose of 600mg AK120 or placebo is administered subcutaneously to healthy subjects
  Arms: Part 1: 600 mg cohort
Drug: AK120 or placebo- Part 2- Cohort 1 — Multiple low doses of AK120 or placebo are administered subcutaneously as a weekly dose for a total of four doses to subjects with moderate-to-severe atopic dermatitis
  Arms: Part 2: low dose cohort
Drug: AK120 or placebo- Part 2- Cohort 2 — Multiple medium doses of AK120 or placebo are administered subcutaneously as a weekly dose for a total of four doses to subjects with moderate-to-severe atopic dermatitis
  Arms: Part 2: medium dose cohort
Drug: AK120 or placebo- Part 2- Cohort 3 — Multiple high doses of AK120 or placebo are administered subcutaneously as a weekly dose for a total of four doses to subjects with moderate-to-severe atopic dermatitis
  Arms: Part 2: high dose cohort
Drug: AK120 or placebo- Part 2- Cohort 4 — Multiple high doses of AK120 or placebo are administered subcutaneously as a bi-weekly dose for a total of three doses to subjects with moderate-to-severe atopic dermatitis.
  Arms: Part 2: Loading dose cohort

SUMMARY:
A dose escalation, first-in-human study evaluating the safety, tolerability, pharmacokinetics, pharmacodynamics and immunogenicity of AK120 in healthy subjects and subjects with moderate- to- severe atopic dermatitis

DETAILED DESCRIPTION:
This is a phase 1, randomized, two-part, double-blind, placebo-controlled, dose-escalation, first-in-human study evaluating the safety, tolerability, pharmacokinetics, pharmacodynamics and immunogenicity of AK120 in healthy subjects (part 1, single ascending dose) and subjects with moderate- to- severe atopic dermatitis(part 2, multiple ascending dose)

ELIGIBILITY:
Major Inclusion Criteria:

Subjects must meet all the following inclusion criteria (as applicable) to be eligible for participation in this study:

Part 1:

1. Willing and able to understand and sign an Informed Consent Form (ICF).
2. Women or men between 18 and 55 years of age, inclusive, at screening.
3. Must have a calculated body mass index within 18.0 to 30.0 kg/m2 (inclusive) at screening, and a total body weight ≥50 kg for men or ≥45 kg for women at screening and Day -1 before randomization.
4. Women of childbearing potential who are sexually active must use one of the permitted methods of contraception from screening until at least 180 days after dosing of study medication.
5. Non-sterilized male subjects who are sexually active with a female partner of childbearing potential must use an effective method of contraception from Day 1 through 180 days after dosing of study medication.
6. Must, in the opinion of the Investigator, be in good general health based upon medical history, physical examination (including vital signs), and 12-lead ECG; and clinical laboratory tests

Part 2:

1. Male or female, aged 18 to 65 years (inclusive) at time of Screening.
2. Chronic atopic dermatitis (AD) diagnosed by the revised Hanifin and Rajka criteria that has been present for at least 1 year before the Screening visit.
3. EASI score ≥12 at the screening and baseline visits.
4. IGA score ≥3 at the screening and baseline visits.
5. BSA of AD involvement ≥10% at the screening and baseline visits.
6. History of an inadequate response or medically inappropriate use of topical drug treatment, in the judgment of the Investigator, to AD treatment with a topical regimen of corticosteroids, phosphodiesterase inhibitors or calcineurin inhibitors or with phototherapy within 6 months of the Screening visit.
7. Subjects must be applying stable doses of an additive-free, basic bland emollient twice daily for at least 7 days before the baseline visit.

Major Exclusion Criteria:

Subjects who meet any of the following exclusion criteria will not be enrolled in this study:

Part 1:

1. Clinically significant clinical safety laboratory result, or blood pressure or electrocardiogram (ECG) abnormalities.
2. Current acute infection or history of acute infection within 7 days prior to receipt of the study drug.
3. Have a recent history of conjunctivitis or keratitis within 6 months prior to screening.
4. History or complications of tuberculosis, or evidence of latent tuberculosis by QuantiFERON®-TB Gold screening.
5. Are positive for hepatitis B surface antigen, hepatitis C antibodies, or human immunodeficiency virus (HIV) at screening.

Part 2:

1. The washout period for prior drug therapy (eg. corticosteroids, immunosuppressive/immunomodulating, biologics, phototherapy, Chinese medicine，anti-infective agents) is inadequate.
2. Any medical or psychiatric condition, laboratory or ECG parameter which, in the opinion of the Investigator or the Sponsor's medical monitor, would place the subject at risk, interfere with participation in the study, or interfere with the interpretation of study results.
3. History of exposure to active TB, and/or history or current evidence of TB infection; and/or Chest X-ray showed old TB lesions at Screening or within 3 months before the Screening visit ..
4. Positive results at Screening for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) or hepatitis C antibody with positive hepatitis C virus (HCV) RNA polymerase chain reaction; positive HIV serology at screening.
5. Any history of vernal keratoconjunctivitis (VKC) and atopic keratoconjunctivitis (AKC) within 6 months before the baseline visit.
6. History of clinical parasite infection, recent or planned travel to an area with endemic parasite infection within 6 months before the Screening visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Adverse events(AEs)/serious adverse events(SAEs) | From signing of informed consent through through 12 weeks post-dose
  Incidence of treatment emergent adverse events(AEs)/serious adverse events(SAEs)

SECONDARY OUTCOMES:
Thymus and activation regulated chemokine (TARC)/Chemokine Ligand 17(CCL17) | From baseline through 12 weeks post-dose
  Change from baseline in serum levels of thymus activation and regulated chemokine (TARC)/Chemokine Ligand 17 (CCL17) in serum
Maximum observed serum concentration (Cmax) | From baseline through 12 weeks post-dose
  Maximum observed serum concentration (Cmax) of AK120
Area under the concentration-time curve (AUC) | From baseline through 12 weeks postdose
  Area under the concentration-time curve (AUC) of serum concentration of AK120
Anti-drug antibodies(ADAs) | From baseline through 12 weeks postdose
  Number and percentage of subjects who develop detectable anti-drug antibodies(ADAs)
Investigator global assessment (IGA) (part 2) | From baseline through 12 weeks postdose
  The proportion of subjects with Investigator global assessment (IGA) 0 to 1 and subjects with IGA reduction from baseline of ≥ 2-point.
  IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a static 6-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe；5 = very severe) based on erythema and papulation/infiltration.
Pruritus-Numeric Rating Scale (P-NRS) (part 2) | From baseline through 12 weeks postdose
  The proportion of subjects with Pruritus-Numeric Rating Scale (P-NRS) improvement (reduction) from baseline of ≥ 3-point.
  Pruritus NRS is an assessment tool that is used to report the intensity of participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable])
Change from baseline in Eczema Area and Severity Index (EASI) score(part 2) | From baseline through 12 weeks postdose
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD). The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Change from baseline in body surface area (BSA) of AD involvement. (part 2) | From baseline through 12 weeks postdose
  Body surface area determined by palm method where 1 palm is equivalent to 1%. Total body surface area ranges from 1% to 100%, with the higher body surface area reflecting the worse severity of AD.

CONTACTS AND LOCATIONS:
Locations (13):
- Australia (6):
  - Emeritus Sydney, Botany, New South Wales
  - Emeritus Melbourne, Camberwell, Victoria
  - CMAX Clinical Research, Adelaide
  - Sinclair Dermatology, East Melbourne
  - Peninsula Specialist Centre, Kippa-Ring
  - Scientia Clinical Research Ltd, Randwick
- New Zealand (7):
  - Southern Clinical Trials - Waitemata, Birkenhead, Auckland
  - Optimal Clinical Trials, Auckland
  - Christchurch Clinical Studies Trust, Christchurch
  - Southern Clinical Trials - Christchurch, Christchurch
  - P3 Research Hawkes Bay, Havelock North
  - P3 Research Tauranga, Tauranga
  - P3 Research Wellington, Wellington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wynne CJ, Cole A, Lemech C, Wang G, Zhang Y, Chen B, Wang M, Li B, Xia M, Sinclair R. Safety, Pharmacokinetics and Preliminary Efficacy of IL4-Ralpha Monoclonal Antibody AK120 in Both Healthy and Atopic Dermatitis Subjects: A Phase I, Randomized, Two-Part, Double-Blind, Placebo-Controlled, Dose-Escalation, First-In-Human Clinical Study. Dermatol Ther (Heidelb). 2023 Oct;13(10):2357-2373. doi: 10.1007/s13555-023-01010-1. Epub 2023 Sep 5. PMID 37668898